CLINICAL TRIAL: NCT03401255
Title: Prospective Multicentric Study Estimating the Interest of a Vaginal Swab in Detection of Placental Alpha-Microglobulin-1 (Partosure®) in the Prediction of Preterm Birth
Brief Title: Interest of a Vaginal Swab in Detection of Placental Alpha-Microglobulin-1 in the Prediction of Preterm Birth
Acronym: MAPOSURE
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0247
Record Dates: First submitted 2018-01-03; First posted 2018-01-17 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Preterm Labor; Preterm Birth
Keywords: Placental alpha microglobulin-1; PAMG-1; preterm labor; preterm delivery; preterm birth; cervical length; transvaginal ultrasound; corticosteroid
MeSH Terms: conditions — Obstetric Labor, Premature; Premature Birth

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — To perform the analysis, a sample of cervicovaginal secretions is collected using a vaginal swab provided in the PAMG-1 Detection Test Kit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Partosure test — To perform the analysis, a sample of cervicovaginal secretions is collected using a vaginal swab provided in the PAMG-1 Detection Test Kit.After removing the swab from its packaging, hold the swab in the middle of the stem and carefully insert the end of the swab into the vagina over a length of 5-7cm (using a speculum). Is not necessary for sampling), when the patient is lying down.Remove the swab from the vagina after 30 seconds. Once the swab has been removed, immediately place the end in the solvent vial provided for this purpose, then rinse the swab by repeating several rotations for 30 seconds. The strip is removed as soon as two bands are clearly visible in the test area, or after 5 minutes.Two bands in the test area indicate a positive result, while a line in the test area indicates a negative result. It is not recommended to read or interpret results beyond 10 minutes of immersion.

SUMMARY:
Preterm labor is the first cause of hospitalization during the pregnancy, and at the origin of more than 60 000 births before 37 weeks of amenorrhea every year in France. It is however difficult to predict if a patient consulting in emergencies with symptoms of preterm labor, will give birth prematurely or not. Current diagnostic tools to identify patients with high risk of premature delivery in 7 days are insufficient because of their low positive predictive value. Yet the neonatal complications in case of premature delivery are important, with respiratory distress syndrome, hyaline membrane disease, necrotizing enterocolitis, intraventricular hemorrhage and post-natal death. Recent studies suggested that the detection of the placental alpha microglobulin 1 (PAMG-1) in the vaginal secretions, by Partosure® test at the women presenting symptoms of preterm labor with intact membranes would indicate that a premature spontaneous delivery could arise in 7 days with a good positive predictive value.The test is interesting all the more as the repetition of the prenatal cures of corticosteroids, aiming at the fetal lung maturation, is this day more recommended and as the beneficial effect takes place within 24 hours in 7 days following their administration. It seems thus essential to make studies to specify the interest of this test at the patients presenting a preterm labor. This study aims at estimating the diagnostic performance of the test of detection of PAMG-1 in the prediction of a delivery in 7 days, at the patients presenting symptoms of preterm labor.

DETAILED DESCRIPTION:
Preterm labor is the first cause of hospitalization during the pregnancy and complicates of a premature delivery in about 30 % of the cases during single pregnancy. It is about a clinical situation arising between 22 and 36 amenorrhea weeks (SA) + 6 days, which are observed the cervical modifications and the uterine contractions confirmed by an ultrasound measure with cervical length ≤25mm.The main complication of the threat premature delivery (MAP) is the premature birth, which is an essential factor of perinatal morbidity and is the second cause of death before the age of 5 years. The measure of cervical length with ultrasound and the detection of the fetal fibronectin were estimated to identify the patients with risk of spontaneous premature delivery, however their capacity to discriminate these patients is insufficient (predictive value is positive of 20 %). It thus seems necessary to find a diagnostic alternative more relevant.The prenatal corticosteroid therapy is recommended for all the patients at risk of premature delivery in 7 days between 24 and 34 SA. Indeed the maximal profit of corticoids arises when the delivery occurs between 12 hours and 7 days following their administration, with a significant reduction in neonatal period the hyaline membrane diseases (50 %), intraventricular hemorrhage, necrotizing enterocolitis and deaths (40 %). Thus corticosteroids establishes the most important treatment in the prematurity.However, the beneficial effect of the corticosteroid therapy decreases if the birth arises beyond 7 days after the administration. So the efficiency of a complete cure of corticoids in the prevention of the neonatal respiratory morbidity is in connection with deadline between the administration and the delivery. The challenge consists in administering the cure of corticoids in 7 days preceding the birth to benefit from the maximal neonatal profit. Besides, the repetition of the cures of corticoids could be responsible for noxious effects on the future of the future adult by distorting the growth of the child and its cognitive future, by increasing the risk of obesity or insulin resistance, as well as the cardiovascular risk in the adulthood.The capacity to discriminate between the patients who are going to give birth prematurely in 7 days so answers a double objective: allow the implementation of an effective and beneficial preventive treatment for the newborn child and avoid treatments and inconvenient hospitalizations, generators of unwanted effects and useless spending.A recent study estimates the interest of an interesting molecule, the placental alpha microglobulin 1 (PAMG-1), in this diagnostic approach. She concludes that the detection of PAMG-1 by a vaginal taking is the best test to predict spontaneous delivery in 7 days compared with the measure of the cervical length by transvaginal ultrasound and the test of fetal fibronectin. If the performance of the test is validated by the study, the coverage of the patients would be optimized with less frequent and less long hospitalizations, as well as a decrease of treatments pointlessly prescribed at the patients not giving birth finally prematurely (tocolytics, corticoids). For those giving birth prematurely, corticoids could be administered for an optimal deadline to obtain the maximal profit for the newborn child.

ELIGIBILITY:
Inclusion Criteria:

* patients presenting for emergency obstetrical care with signs suggestive of preterm labor
* single pregnancy
* gestational age between 24 + 0 and 33SA + 6 weeks of gestation
* cervical length ≤ 25mm measurement on transvaginal ultrasound with or without uterine contraction
* informed consent
* consenting to be part of the trial

Exclusion Criteria:

* < 18 years old or patient under guardianship / curators
* multiple pregnancy
* gestational term less than 24 SA or greater than or equal to 34 SA
* heavy vaginal bleeding- antecedent of conisation
* uterine malformation ( bicervical-bicorn uterus, unicervical bicorn uterus, unicorn uterus, septate uterus)
* Cervical dilatation >3 cm.
* cervical length with transvaginal ultrasound >25mm
* presence of a hydramnios with a superior amniotic fluid index 25
* premature rupture of manifest membranes (PROM)
* clinical or biological chorioamnionitis
* hooping cervical
* intercurrent obstetric pathology that can induce premature birth
* patient hospitalized for more than 24 hours in another hospital or service for preterm labor diagnosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting symptoms of preterm labor
Sampling Method: Non-Probability Sample
Enrollment: 341 (Actual)
Dates: Start 2018-02-28 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
diagnostic performance of detection test of PAMG-1 for the prediction of imminent spontaneous preterm delivery within 7 days in patients presenting with symptoms of preterm labor | time to delivery
  The diagnostic performance of the test will be evaluated by estimating its specificity.

SECONDARY OUTCOMES:
sensitivity of detection test of PAMG-1 | time to delivery
  To evaluate the diagnostic performance (sensitivity) of detection test of PAMG-1 for the prediction of imminent spontaneous preterm delivery within 7 days in patients presenting with symptoms of preterm labor.
positive predictive of detection value test of PAMG-1 | time to delivery
  : To evaluate the diagnostic performance (positive predictive value) of detection test of PAMG-1 for the prediction of imminent spontaneous preterm delivery within 7 days in patients presenting with symptoms of preterm labor.
negative predictive of detection value test of PAMG-1 | time to delivery
  To evaluate the diagnostic performance (negative predictive value) of detection test of PAMG-1 for the prediction of imminent spontaneous preterm delivery within 7 days in patients presenting with symptoms of preterm labor.
diagnostic performance of detection test of PAMG-1 in the prediction of imminent spontaneous preterm delivery within 48 hours in patients presenting with symptoms of preterm labor. | time to delivery
  The result of PAMG-1 test at the time of hospitalization (positive / negative), interval between hospitalization and delivery +/- 48 hours will be collected
cervical length at inclusion | within 48 hours after delivery
  Delivery within 48 hours if cervical length is less than 15 mm, 15-19 mm and 20-25 mm at the time of inclusion and delivery within 48 hours if gestational age is between 24 weeks of amenorrhea (SA) and 27 SA + 6, 28 SA and 31 SA + 6, 32 SA and 33 SA + 6 at the time of inclusion and the result of PAMG-1 test will be recorded.
cervical length at inclusion | within 7days after delivery
  Delivery within 7 days if cervical length is less than 15 mm, 15-19 mm and 20-25 mm at the time of inclusion and delivery within 7 days if gestational age is between 24 SA and 27 SA + 6, 28 SA and 31 SA + 6, 32 SA and 33 SA + 6 at the time of inclusion and the result of PAMG-1 test will be recorded.
gestational age at inclusion | within 48hours after delivery
  Delivery within 48 hours if cervical length is less than 15 mm, 15-19 mm and 20-25 mm at the time of inclusion and delivery within 48 hours if gestational age is between 24 SA and 27 SA + 6, 28 SA and 31 SA + 6, 32 SA and 33 SA + 6 at the time of inclusion and the result of PAMG-1 test will be recorded.
gestational age at inclusion | 7 days within after delivery
  Delivery within 7 days if cervical length is less than 15 mm, 15-19 mm and 20-25 mm at the time of inclusion and delivery within 7 days if gestational age is between 24 SA and 27 SA + 6, 28 SA and 31 SA + 6, 32 SA and 33 SA + 6 at the time of inclusion and the result of PAMG-1 test will be recorded.
False positives. | time to delivery
  evaluate factors associated for patients with a positive test who did not give birth within 7 days Gestational age less than 34 weeks and 37 weeks at the time of birth.
hospital stays | time to delivery
  Economic impact evaluation
PAMG-1 tests consumption | time to delivery
  Economic impact evaluation
corticosteroid treatments consumption | time to delivery
  Economic impact evaluation
tocolytic treatments consumption | time to delivery
  Economic impact evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Dochez, PH, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - La Roche-sur-yon University Hospital, La Roche-sur-Yon
  - Nantes University Hospital, Nantes

REFERENCES:
- [Derived] Marie E, Ducarme G, Boivin M, Badon V, Pelerin H, Le Thuaut A, Lamoureux Z, Riche VP, Winer N, Thubert T, Dochez V. The value of a vaginal sample for detecting PAMG-1 (Partosure(R)) in women with a threatened preterm delivery (the MAPOSURE Study): protocol for a multicenter prospective study. BMC Pregnancy Childbirth. 2020 Aug 3;20(1):442. doi: 10.1186/s12884-020-03129-x. PMID 32746802